CLINICAL TRIAL: NCT01107691
Title: Resistance Training Energy Balance & Weight Management
Brief Title: Comparison of 1 vs 3 Sets of Resistance Training on Muscular Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Washburn, Associate Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSCL17623; NIDDKRO180832 (Other Grant/Funding Number: National Institues of Health)
Record Dates: First submitted 2010-03-26; First posted 2010-04-21 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: resistance and weight loss training
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resistance training (Experimental): 1 set of progressive resistance training per session
  Interventions: Other: Amount of resistance offered in training
- 3 sets per session (Experimental): 3 sets of progressive resistance training per session
  Interventions: Other: Amount of resistance offered in training
- Control (No Intervention): Non exercise control group

INTERVENTIONS:
Other: Amount of resistance offered in training — to determine the impact of the volume (1 vs. 3 sets) of a progressive resistance training protocol for inducing muscular hypertrophy
  Arms: 3 sets per session; Resistance training

SUMMARY:
This study is designed to investigate the effects of two levels of resistance weight training on body composition, energy expenditure, and energy intake in men and women. The weight training will take about one hour to complete. Participants will perform the training 3 days per week for 9 months in a private exercise room equipped with state of the art equipment and a personal trainer to help guide you through the exercises.

The project lasts 21 months total with one follow-up visit 1-year from your last training date. You will be required to stay in the Lawrence area and train 3 day/week over the summer & holidays.

DETAILED DESCRIPTION:
We propose to conduct a randomized controlled efficacy trial (RT-1 set vs. RT-3 sets vs. non exercise control) to evaluate the potential for a longer intervention (9 months RT with body composition assessments 1 yr post RT completion) with a higher volume of RT (3 sets) to enhance the effects on body composition and energy expenditure observed in the pilot, and to determine the impact of the 2 levels of RT on free-living energy balance (expenditure by doubly labeled water and intake by digital photography and 24-hr recalls). This investigation will be conducted in a sample of healthy, normal and overweight, sedentary, young adult men and women; a group at high risk for development of overweight and obesity. The specific aims of this project are to determine the impact of the volume (1 vs. 3 sets) of a progressive RT protocol for inducing muscular hypertrophy, as recommended by the American College of Sports Medicine, on body weight and body composition (fat mass, fat-free mass (FFM), % body fat) and energy balance. Our results will provide information relative to the minimum volume of RT that may be associated with body weight/fat gain which may inform the development of guidelines for RT to prevent weight gain or to alter body composition. If RT has a favorable impact on energy balance and body composition, it may provide an attractive alternative to aerobic exercise for weight management for busy young adults, as RT requires minimal time, and no need to change clothes or shower (i.e. minimal or no sweating).

ELIGIBILITY:
Inclusion Criteria:

* BMI 22-<30
* 18- 30 years old
* sedentary
* no medications
* weight stable for at least 3 months

Exclusion Criteria:

* Tobacco/Drug user
* metabolism altering medication
* gain/lost 10lbs in the last 3 months
* current exerciser

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2009-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Body Composition | 21 Months
  Changes in body composition will be evaluated by measuring the change in percent body fat, total fat mass, and total lean mass by dual energy x-ray absorptiometry (DEXA).

SECONDARY OUTCOMES:
Resting Metabolic Rate | 9 months
  Resting metabolic rate as measured by indirect calorimetry as kcal/day will be evaluated. Also, substrate oxidation (fat and carbohydrate oxidation) will be evaluated at these time points.
Muscular Strength | 9 months
  One rep max strength will be measured on the chest and leg press.
Daily Energy Expenditure | 9 months
  Total daily energy expenditure over a 14 day period will be measured using doubly labeled water.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Washburn, PhD, Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States